CLINICAL TRIAL: NCT01301261
Title: The Effect of Sugammadex on Hemodynamics, Oxygenation, End-tidal CO2, Entropy and Bispectral Index Intraoperatively Without Steroid Neuromuscular Blocker
Brief Title: Sugammadex: Effect on the Awareness Monitoring and Hemodynamics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Argyro Fassoulaki, MD, PhD, DEAA, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Σ-150/03-08-10
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Surgical Procedure, Unspecified
Keywords: Sugammadex; entropy; bispectral index; blood pressure; heart rate; oxygenation; end-tidal CO2; hemodynamics; general anesthesia
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- sugammadex 2 mg/kg (Active Comparator): 2 mg/kg of sugammadex are given when a response of two counts of train of four are present
  Interventions: Drug: sugammadex
- 4 mg/kg of sugammadex (Active Comparator): 4 mg/kg of sugammadex are given when a posttetanic count 1-3 appears
  Interventions: Drug: Sugammadex 4 mg/kg
- Sugammadex 16 mg/kg (Active Comparator): Sugammadex 16 mg/kg are given three minutes after the injection of cis-atracurium
  Interventions: Drug: Sugammadex 16mg/kg

INTERVENTIONS:
Drug: sugammadex — Sugammadex 2 mg/kg when a two count of train of four appears
  Arms: sugammadex 2 mg/kg
Drug: Sugammadex 4 mg/kg — Sugammadex 4 mg/kg are given when a posttetanic count 1-3 appears
  Arms: 4 mg/kg of sugammadex
Drug: Sugammadex 16mg/kg — Sugammadex 16 mg/kg three minutes after the injection of cis-atracurium
  Arms: Sugammadex 16 mg/kg

SUMMARY:
Sugammadex is used to reverse the neuromuscular blocking effect of steroid neuromuscular blockers. Its cardiovascular effects and effect on brain cortex, if any, may be associated to the reversal of the neuromuscular block. The aim of the study was to investigate the pure effects of sugammadex in the absence of the agonist.

DETAILED DESCRIPTION:
Three groups of patients undergoing elective major surgery and given cis-atracurium for muscle relaxation are studied.

Group 1 receives 2 mg/kg of sugammadex when a count of two of the train of four appears Group 2 receives 4 mg/kg of sugammadex when a posttetanic count 1-3 appears Group 3 receives 16 mg/kg of sugammadex three minutes after administration of cis-atracurium.

Heart rate, arterial blood pressure, oxygen saturation, end-tidal CO2, entropy and bispectral index are recorded every three minutes

ELIGIBILITY:
Inclusion Criteria:

* patients ASA I-III scheduled for elective major surgery
* both sexes

Exclusion Criteria:

* patients hypertensive
* treated with antihypertensive drugs

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Entropy | every three minutes

SECONDARY OUTCOMES:
hemodynamics | every three minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Aretaieio Hospital, Athens, Greece